CLINICAL TRIAL: NCT00299741
Title: A Phase II Study of SU011248 in Men With Advanced Prostate Cancer
Brief Title: Study of SU11248 in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dror Michaelson, MD, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-05-1-0439
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Results first posted 2012-12-13 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Prostate Cancer
Keywords: Sutent; Sunitinib; Bone; Metastatic; Hormone-refractory; Biomarkers
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sunitinib
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 50 mg daily, 4/2 schedule
  Other Names: Sutent

SUMMARY:
* There are nearly 30,000 deaths per year in the United States from prostate cancer, making this a large and important target patient population for new cancer treatments.
* SU011248 is an exciting, new, experimental drug that inhibits a number of proteins, or more specifically receptor tyrosine kinases, in tumor cells. These proteins are active in cellular pathways that are important for development and growth of a variety of different cancers. The targets of SU011248 include the receptors for vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), and others. By blocking the VEGF and PDGF pathways, SU011248 can induce death of the blood vessels that nourish the cancer cells and death of the cancer cells themselves.
* SU011248 has demonstrated significant anti-tumor activity in renal cell carcinoma, gastrointestinal stromal tumors, and other cancers. Its effect against prostate cancer has not been studied to date.
* This study is directed at two populations of men with advanced prostate cancer:

  1. Men with advanced prostate cancer who have a rising PSA despite hormone therapy, but have not yet received any chemotherapy.
  2. Men with metastatic prostate cancer who have received prior chemotherapy (with a docetaxel-based regimen) and have increasing disease following chemotherapy.
* Men in this study will receive SU011248 on a six-week repeating schedule, with four weeks of daily treatment followed by a two-week rest. The goals of the study are:

  1. to determine whether SU011248 is an important therapeutic agent in men with advanced prostate cancer, and
  2. to identify predictive markers of anti-cancer activity within individual subjects that would allow selective treatment of appropriate subjects in the future.

DETAILED DESCRIPTION:
Background: There are nearly 30,000 deaths per year in the United States from prostate cancer, making this a large and important target patient population for new therapeutics. The mainstay of therapy for advanced prostate cancer is androgen deprivation therapy (ADT). Although ADT is effective in the large majority of men with advanced prostate cancer, the favorable response to ADT is only transient. In hormone-refractory, metastatic prostate cancer the only effective systemic treatment is cytotoxic chemotherapy. The median duration of response to standard, taxane-based chemotherapy is approximately six months, and median survival in contemporary studies is only 16-18 months. Thus, there is an urgent need for new therapeutic agents to treat advanced prostate cancer.

SU011248 is an orally administered inhibitor of the vascular endothelial growth factor (VEGF) receptors, platelet-derived growth factor (PDGF) receptor, FLT-3 and c-KIT. SU011248 has demonstrated significant clinical activity in other malignancies, but its activity in prostate cancer has not been studied to date. Clinical trials have demonstrated that SU011248 is generally well tolerated, with mild fatigue and diarrhea the most common adverse effects. Preclinical studies have demonstrated that levels of VEGF and PDGF are elevated in prostate cancer and may correlate with worse outcome. The inhibition of several pathways implicated in prostate cancer progression by SU011248 suggests that it might have significant anti-tumor activity in men with AIPC.

Many of the new, targeted agents are efficacious in only a subset of patients with a particular malignancy, and these subsets may be definable on the basis of specific tumor mutations or patterns of gene expression. Identification of reliable predictive methods is crucial in moving forward with targeted therapies, and we believe that exploratory clinical trials such as this one should incorporate assays designed to address this issue.

Objective/Hypothesis: The objective of this proposal is to determine whether SU011248 is an effective treatment in two cohorts of men with advanced prostate cancer: men with androgen-independent prostate cancer (AIPC) who have not been treated with chemotherapy (Group A), and men with taxane-refractory, metastatic disease (Group B). We hypothesize that specific serum biomarkers and tumor mutations may predict response and may allow optimal subject selection in the future.

Specific Aims: (1) To evaluate the efficacy and safety of SU011248 in men with chemo-naïve AIPC, (2) to evaluate the efficacy and safety of SU011248 in men with metastatic, taxane-resistant AIPC, (3) to measure serum biomarkers in men with AIPC prior to and following treatment with SU011248 and correlate these markers with clinical response, and (4) to mutational analysis from tumor specimens of men with metastatic prostate cancer treated with SU011248 and correlate with clinical response.

Study Design: We will conduct a phase II clinical trial in two groups of subjects: men with AIPC who have not yet developed overt metastases (Group A), and men with taxane-refractory, metastatic disease (Group B). Men in both groups will receive single-agent SU011248 on a six-week repeating schedule, with four weeks of daily treatment followed by a two-week rest. The primary endpoint will be PSA response rate. Secondary endpoints will include time to disease progression, objective response rate, and safety parameters. Eligibility for this study will require signed informed consent, adenocarcinoma of the prostate, documented PSA progression despite ADT, reasonable functional status, resolution of toxic effects from prior treatments, and acceptable bone marrow, hepatic, renal and cardiac function. A Simon's two-stage design will be employed to allow early termination for lack of efficacy. Ultimately, 30 patients will be enrolled in each group, for a total of 60 patients. A defined program of history and physical examinations, radiographic studies, and laboratory tests including PSA will be carried out to determine the efficacy and safety of SU011248 in this patient population.

All subjects will have blood and urine collected for research purposes, and men in Group B will have tumor biopsy prior to enrollment. Translational studies aimed at identifying specific biomarkers in the blood will include analysis of serum cytokine levels including VEGF and others, circulating endothelial cells and endothelial precursors, white blood cell differential, and bone turnover markers. Tumor samples will be analyzed for the presence of predictive tumor mutations.

Relevance: Our ultimate goals are to determine whether SU011248 is an important therapeutic agent in men with advanced prostate cancer, and to identify predictive markers of anti-cancer activity within individual subjects that would allow selective treatment of appropriate subjects in the future. The data obtained should also contribute to our general understanding of serum biomarkers and genetic changes in advanced prostate cancer. Positive results of our trial would lead to expanded, multi-center trials of SU011248 in men with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent indicating that the subject has been informed of all pertinent aspects of the trial.
* Adenocarcinoma of the prostate
* Male subjects, 18 years of age or older
* Life expectancy of > 12 weeks
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy or surgical procedure to National Cancer Institute Common Toxicity Criteria Adverse Event (NCI CTCAE) grade <1
* Surgical or ongoing chemical castration
* Androgen-independent disease, defined as progressive disease despite surgical or ongoing chemical castration. See section 8.2.3 for definition of progressive disease.
* Eastern Cooperative Oncology Group performance status of 0, 1 or 2
* Adequate bone marrow reserve:

  * Neutrophil count > 1,500/ul
  * Platelet count > 75,000/ul
* Adequate hepatic function:

  * Serum bilirubin < 1.5 x upper limit of normal
  * Asparate aminotransferase and alanine aminotransferase < 2.5 x upper limit of normal
* Adequate renal function, with serum creatinine < 2 x upper limit of normal
* Prostate Specific Antigen (PSA) > 5.0 ng/mL, based on PSA Working Group Criteria
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

For Group A only:

· No prior treatment for prostate cancer with cytotoxic chemotherapy

For Group B only:

* Radiographic evidence of metastatic prostate cancer
* One prior docetaxel-based chemotherapy regimen, minimum of two cycles
* Disease progression during treatment with docetaxel, or within 60 days of receiving docetaxel

Exclusion Criteria:

* Small cell carcinoma of the prostate
* Treatment with extensive external beam radiation therapy or radionuclide therapy within six weeks of study entry. Palliative radiation involving less than 20% of bone marrow reserves must have been completed within four weeks of entry.
* Any of the following within the prior 6 months: unstable angina, myocardial infarction, symptomatic congestive heart failure or cerebrovascular accident
* Receipt of any investigational anti-cancer agent within 4 weeks of the study
* NCI CTCAE grade 3 hemorrhage < 4 weeks of starting study treatment
* Uncontrolled hypertension
* Prolongation of the QTc interval to > 450 msec
* Other serious acute or chronic medical or psychiatric condition that may increase the risk associated with study participation, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Michaelson, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel-Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Dror Michaelson M, Regan MM, Oh WK, Kaufman DS, Olivier K, Michaelson SZ, Spicer B, Gurski C, Kantoff PW, Smith MR. Phase II study of sunitinib in men with advanced prostate cancer. Ann Oncol. 2009 May;20(5):913-20. doi: 10.1093/annonc/mdp111. PMID 19403935
- [Derived] Saylor PJ, Mahmood U, Kunawudhi A, Smith MR, Palmer EL, Michaelson MD. Multitargeted tyrosine kinase inhibition produces discordant changes between 99mTc-MDP bone scans and other disease biomarkers: analysis of a phase II study of sunitinib for metastatic castration-resistant prostate cancer. J Nucl Med. 2012 Nov;53(11):1670-5. doi: 10.2967/jnumed.112.105007. Epub 2012 Sep 14. PMID 22984218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients identified from routine care in oncology clinic
Groups:
- Metastatic Prostate Cancer Treated With Sunitinib: Sunitinib administered orally at a dosage of 37.5 mg once daily
Period: Overall Study
Arm/Group | Metastatic Prostate Cancer Treated With Sunitinib
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Metastatic Prostate Cancer Treated With Sunitinib: Sunitinib
Arm/Group | Metastatic Prostate Cancer Treated With Sunitinib
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: The Number of Men With Advanced Prostate Cancer Treated With Sunitinib Who Have a Prostate Specific Antigen (PSA) Response
Description: Prostate specific antigen (PSA) responses, defined as the number of men who exhibit PSA decline of at least 50% that is confirmed by a second PSA value 4 or more weeks later (PSA Working Group I Criteria)
Time Frame: were followed until disease progression, an average of 12 weeks
Population: All participants analyzed
Measure: Number; unit: participants
Arm/Group | Metastatic Prostate Cancer Treated With Sunitinib
Number analyzed (Participants) | 36
participants | 2

2. Secondary Outcome: Objective Responses, Defined as the Number of Participants With Complete or Partial Response
Description: The response rate is defined by Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions as assessed by radiographic evaluation. Complete response(CR): disappearance of all target lesions; Partial response(PR): >=30% decrease in the sum of the longest diameter of target lesions; Overall response = CR + PR.
Time Frame: Participants were followed until the time of disease progression, an average of 12 weeks
Measure: Number; unit: participants
Arm/Group | Metastatic Prostate Cancer Treated With Sunitinib
Number analyzed (Participants) | 36
participants | 1

ADVERSE EVENTS:
Time Frame: Throughout treatment period
Arm/Group | Metastatic Prostate Cancer Treated With Sunitinib
Serious Adverse Events (participants affected / at risk) | 25/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Prostate Cancer Treated With Sunitinib (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Leukocytes (Blood and lymphatic system disorders) | 6 (6)
Neutrophils (Blood and lymphatic system disorders) | 5 (5)
Platelets (Blood and lymphatic system disorders) | 4 (4)
ALT/AST elevation (Hepatobiliary disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (1)
Hyponatremia (Renal and urinary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 5 (5)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Lower GI hemorrhage (Gastrointestinal disorders) | 1 (1)
Neuropathy - sensory (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Thrombosis/Embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No